CLINICAL TRIAL: NCT06333379
Title: Non-Invasive Detection of Aspergillosis in Ventilated Patients: Galactomannan Analysis in Exhaled Breath
Brief Title: Aspergillosis Detection Via EBC-GM in Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, chief physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: SichuanPPHLC04; 2020LY01 (Other Grant/Funding Number: Sichuan Provincial People's Hospital)
Record Dates: First submitted 2024-03-18; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Bronchoalveolar Lavage Fluid; Sensitivity and Specificity; Critical Illness; Respiration Failure; Respiratory Fungal Infection; Exhaled Breath Condensate; Aspergillosis, Invasive Pulmonary
Keywords: Exhaled breath condensation; Bronchoalvelar lavage fluid; Galactomannan; Invasive Pulmonary Aspergillosis; Non-invasive diagosis
MeSH Terms: conditions — Hypersensitivity; Critical Illness; Respiratory Insufficiency; Invasive Pulmonary Aspergillosis | interventions — Floors and Floorcoverings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The investigators collected bronchoalveolar lavage fluid (BALF) and exhaled breath condensate (EBC) specimens from all patients for GM testing. One of the BALF specimens also needed to be sent for culture and macrogenomic sequencing in Invasive Aspertillosis Pneumonia(IPA) group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPA group: Investigators enrolled patients who meet diagnostic criteria for IPA according to EORTC/MSG: new exudative lung lesions unresponsive to antimicrobial therapy; positive Aspergillus on LRT and/or BALF microscopy cultures, positive BALF GM and positive BALF NGS results for Aspergillus. Investigators will test and compare the EBC-GM and BALF-GM levels in these patients.
  Interventions: Other: Compare the levels of Galactomannan (GM) levels in exhaled breath condensate (EBC) and BALF
- control group: Investigators enrolled patients who were mechanically ventilated patients without Aspergillus infection or colonization. BALF and EBC samples from the same patients were collected less than 4 hours apart, and BALF samples were used for NGS and microbiological cultures. Investigators will test and compare the EBC-GM and BALF-GM levels in these patients.
  Interventions: Other: Compare the levels of Galactomannan (GM) levels in exhaled breath condensate (EBC) and BALF

INTERVENTIONS:
Other: Compare the levels of Galactomannan (GM) levels in exhaled breath condensate (EBC) and BALF — Investigators tested EBC-GM levels and BALF-GM levels in patients with confirmed IPA to compare the diagnostic value of EBC-GM versus BALF-GM.

SUMMARY:
Brief Research Proposal: Non-Invasive Detection of Invasive Pulmonary Aspergillosis in ICU Patients Background: Invasive Pulmonary Aspergillosis (IPA) is a critical threat to patients in ICUs, especially those undergoing mechanical ventilation. Traditional diagnostic methods are invasive and carry risks. This study proposes a non-invasive, innovative approach utilizing galactomannan (GM) analysis in Exhaled Breath Condensate (EBC) for early IPA detection.

Objective: To evaluate the diagnostic accuracy of measuring GM levels in EBC for detecting IPA in mechanically ventilated patients, comparing it against the conventional Bronchoalveolar Lavage Fluid (BALF)-GM measurements.

Methods: A clinical trial will be conducted with 75 mechanically ventilated patients suspected of having IPA. The study will compare the effectiveness of EBC-GM levels against BALF-GM levels in diagnosing IPA, focusing on sensitivity, specificity, and diagnostic accuracy. The novel, self-designed EBC collection device will facilitate the safe and efficient collection of EBC from patients.

Expected Outcomes:

Validation of EBC-GM Diagnostic Accuracy: Anticipate demonstrating that EBC-GM levels provide a comparable diagnostic accuracy to BALF-GM, establishing a non-invasive, safer alternative for IPA detection.

Implementation of a Non-Invasive Diagnostic Tool: The study aims to introduce a non-invasive diagnostic approach that can potentially replace more risky, invasive methods, improving patient care in ICUs.

Contribution to Clinical Practice: By providing a new method for early and safer detection of IPA, the study is expected to influence clinical guidelines and practices in the management of critically ill, ventilated patients.

Significance: This research has the potential to revolutionize the diagnosis of fungal infections in critically ill patients by offering a non-invasive, accurate, and safer diagnostic tool, thereby improving patient outcomes and reducing the risks associated with invasive diagnostic procedures.

DETAILED DESCRIPTION:
Research Proposal: Advancing the Diagnosis of Invasive Pulmonary Aspergillosis through Exhaled Breath Condensate Analysis in Ventilated Patients Background: Invasive Pulmonary Aspergillosis (IPA) remains a formidable challenge in the management of critically ill, immunocompromised patients, especially those requiring mechanical ventilation in Intensive Care Units (ICUs). The high morbidity and mortality rates associated with IPA underscore the urgent need for early and accurate diagnostic methods. Traditional diagnostic approaches, though effective, are invasive and pose significant risks to already vulnerable patients. This study introduces a novel, non-invasive diagnostic methodology by measuring galactomannan (GM) levels in Exhaled Breath Condensate (EBC), potentially revolutionizing the early detection of IPA.

Objective: To evaluate the effectiveness of a non-invasive diagnostic approach by analyzing galactomannan levels in exhaled breath condensate (EBC) for detecting Invasive Pulmonary Aspergillosis (IPA) in mechanically ventilated ICU patients.

Methods:

Study Design: A prospective clinical trial involving 75 mechanically ventilated patients suspected of having IPA within the Medical Intensive Care Unit (MICU) of a tertiary hospital.

Data Collection: Utilizing a self-designed EBC collection device, EBC samples will be collected from participants and analyzed for GM levels. These will be compared to Bronchoalveolar Lavage Fluid (BALF) GM levels, considered the current gold standard in IPA diagnostics.

Analytical Approach: The study will focus on assessing the diagnostic accuracy of EBC-GM measurements by determining sensitivity, specificity, and overall concordance with BALF-GM levels. The potential enhancement of diagnostic precision with the inclusion of cytokine measurements will also be explored.

Innovation: By leveraging a cutting-edge EBC collection device, this research aims to bypass the complications associated with invasive diagnostic procedures, offering a safer, more patient-friendly alternative. This innovative approach has the potential to significantly impact clinical practices in ICU settings by facilitating early and accurate IPA diagnosis without the need for bronchoscopy.

Expected Outcomes:

Diagnostic Performance: Investigators anticipate demonstrating that EBC-GM levels provide a reliable, non-invasive marker for IPA, with diagnostic accuracy comparable to BALF-GM measurements.

Clinical Impact: The successful validation of EBC-GM as a diagnostic tool for IPA will offer a significant advancement in the management of critically ill patients, reducing the need for invasive procedures and associated risks.

Guideline Integration: Findings from this study are expected to support the integration of EBC-GM analysis into clinical guidelines as a recommended diagnostic approach for IPA in mechanically ventilated patients.

Significance: This research has the potential to transform IPA diagnostics in ICU settings, promoting a shift towards non-invasive, risk-free methods that can lead to earlier detection and improved patient outcomes. By minimizing invasive diagnostic interventions, the study aims to enhance the safety and efficacy of IPA management in critically ill populations.

Ethics and Dissemination: The study adheres to the highest ethical standards, with approval from the institutional review board ensuring the protection and well-being of participants. Results will be actively disseminated through peer-reviewed journals and conference presentations, contributing to global efforts in improving ICU patient care in the context of fungal infections.

ELIGIBILITY:
Inclusion Criteria:

- Age: Between 18 and 85 years old. Antifungal Medication Use: Participants who have not used any antifungal medications within the three months prior to enrollment.

Mechanical Ventilation Status: Patients who have been undergoing mechanical ventilation treatment for more than three days.

Exclusion Criteria:

- Inadequate Clinical Data: Inability to provide reliable diagnostic measurements or insufficient clinical information.

Early Mortality: Patients who die within the first three days of ICU (Intensive Care Unit) admission or during the initial phase of the study.

Pregnancy: To avoid potential confounding effects on immune function and the composition of EBC (Exhaled Breath Condensate), pregnant women are excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators at Sichuan Provincial Hospital study mechanically ventilated adults for Invasive Pulmonary Aspergillosis (IPA) risks. They classify participants into IPA and control groups. IPA patients meet EORTC/MSG criteria, showing new lung lesions, positive Aspergillus cultures in LRT, positive galactomannan in BALF, and supporting BALF NGS evidence. The control group includes ventilated patients without Aspergillus, confirmed by negative cultures and NGS in BALF. The study aims to assess EBC-GM's diagnostic accuracy for IPA, comparing it with BALF-GM for early, non-invasive detection.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of EBC-GM vs. BALF-GM | EBC and BALF samples were collected simultaneously on the day of patient admission.
  The diagnostic accuracy of Galactomannan (EBC-GM) levels in Exhaled Breath Condensate vs. Bronchoalveolar Lavage Fluid (BALF-GM) levels was measured by Receiver Operating Characteristic (ROC) area under the curve (AUC) assessment. Accuracy of Galactomannan (BALF-GM) levels in the diagnosis of Invasive Pulmonary Aspergillosis (IPA).
EBC-GM levels: | The stability of the patients' vital signs was observed within 72 hours to assess the diagnostic accuracy of EBC-GM and BALF-GM.
  Evaluate sensitivity and specificity in differentiating patients with IPA from mechanically ventilated patients with non-aspergillosis infections, and determining the critical value of EBC-GM in the diagnosis of IPA.

SECONDARY OUTCOMES:
Correlation between EBC-GM and BALF-GM levels | Based on samples collected on the same day, followed by 72 hours of observation.
  To assess the correlation between EBC-GM levels and BALF-GM levels in mechanically ventilated IPA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, doctoral, Principal Investigator — Sichuan Provincial People's Hospita
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
This study tests a non-invasive method for detecting Invasive Aspergillosis (IPA) in ICU patients using ventilators. By analyzing galactomannan in exhaled breath, we aim to identify IPA without invasive procedures. Phase 1 involves testing a new breath collection device on rats. Phase 2 applies this device to 75 ICU patients, comparing results with traditional lung fluid tests. Approval from an ethics committee ensures patient safety. Successful outcomes could lead to safer IPA diagnosis, enhancing treatment and reducing risks associated with current methods.

REFERENCES:
- [Derived] Tang X, Yang L, Zhang R, Fang H, Tang H, Xie Q, Wang H, Chen L, Yang Y. Non-invasive detection of Aspergillosis in ventilated patients: Galactomannan analysis in exhaled breath. Diagn Microbiol Infect Dis. 2024 Sep;110(1):116420. doi: 10.1016/j.diagmicrobio.2024.116420. Epub 2024 Jun 29. PMID 38954860

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT06333379/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT06333379/ICF_001.pdf